CLINICAL TRIAL: NCT01039519
Title: A Non-randomized, Open Label, Multi-center Phase 2 Study Evaluating the Efficacy and Safety of STA-9090 in Patients With Metastatic and/or Unresectable GIST Resistant or Refractory to Prior Systemic Treatments Including Imatinib and Sunitinib
Brief Title: A Study Evaluating STA-9090 in Patients With Metastatic and/or Unresectable Gastrointestinal Stromal Tumor (GIST)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9090-05
Record Dates: First submitted 2009-12-23; First posted 2009-12-25 (Estimated); Results first posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: G.I. Stromal Tumor; GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — STA 9090

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ganetespib 200 mg/m^2 (Experimental): Ganetespib (STA-9090) 200 mg/m^2 intravenous infusion once weekly for 3 consecutive weeks followed by one week dose free interval (3 weeks on and 1 week off represent a treatment cycle). Treatment continues until disease progression or unacceptable toxicity.
  Interventions: Drug: Ganetespib

INTERVENTIONS:
Drug: Ganetespib — Ganetespib 200 mg/m^2 during an approximately 1-hour infusion once weekly for three consecutive weeks followed by a treatment-free week. Participants who demonstrate acceptable tolerability and objective clinical benefit (defined by at least stable disease or objective response per RECIST) can continue to receive ganetespib until disease progression or appearance of unacceptable toxicity.
  Other Names: STA-9090

SUMMARY:
The purpose of this study is to determine if STA-9090 is effective in the treatment of patients with metastatic and/or unresectable GIST.

DETAILED DESCRIPTION:
Planned:

* Stage 1: 23 patients. If ≥4 patients had clinical benefit, an additional 32 patients were to be enrolled. Up to 3 additional patients with platelet-derived growth factor receptor, alpha polypeptide (PDGFRA) mutation were to be enrolled, regardless of the total study enrollment.
* Stage 2: 55 patients. Progressing to this stage was dependent on Stage 1 results.

Analyzed:

* Stage 1: 27 patients were enrolled and analyzed. The study was not expanded to Stage 2 due to insufficient efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age at the time of study entry
* Must have histologically confirmed metastatic and/or unresectable GIST
* Must have measurable disease on computed tomography or magnetic resonance imaging as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Must have documented failure (due to either progression or intolerance)of at least prior imatinib and sunitinib. Previous administration of other known heat shock protein 90 (Hsp90) inhibitors is permitted
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Must have acceptable laboratory values as defined in the protocol

Exclusion Criteria:

* Known central nervous system metastases
* Major surgery within 4 weeks prior to receiving STA-9090
* Use of any investigational agents within 2 weeks or 6 half-lives of the agent, whichever is shorter prior to receiving STA-9090
* No treatment with chronic immunosuppressants
* Must have otherwise adequate health status as defined in the protocol
* Left ventricular ejection fraction (LVEF) < than or = 50% at baseline
* Baseline corrected QT interval (QTc) > 470 msec
* Pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UCLA Medical Center, Los Angeles, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health and Science University-Knight Cancer Institute, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-one patients were screened; 4 of the 31 were screen failures.
Period: Treatment
Arm/Group | Ganetespib 200 mg/m^2
Started | 27
Completed | 0 (Reason not completed represents reason for terminating treatment.)
Not Completed | 27
Not completed — Progressive disease | 20
Not completed — Treatment failure | 2
Not completed — Adverse Event | 3
Not completed — Physician Decision | 2
Period: Survival Follow-up
Arm/Group | Ganetespib 200 mg/m^2
Started | 27
Completed | 0
Not Completed | 27
Not completed — Death | 23
Not completed — Sponsor decision | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set, which includes participants given at least one dose of study medication.
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 74.94 (22.095)
Height [Mean (Standard Deviation); unit: cm] | 171.57 (10.295)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.863 (0.2909)
Time from Initial Gastrointestinal Stromal Tumor (GIST) Diagnosis to Consent [Mean (Standard Deviation); unit: months] — N = 25 participants
  months | 68.71 (34.699)
Time from Metastatic/Unresectable GIST Diagnosis to Consent [Mean (Standard Deviation); unit: months] — N = 20 participants GIST = gastrointestinal stromal tumor
  months | 46.77 (28.606)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — The ECOG scale is as follows:
  * Grade 0: Fully active, able to carry on all pre-disease activities without restriction;
  * Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  * Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours;
  * Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  * Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or Chair.
  participants
    0 | 14
    1 | 13
Any Prior Exposure to Heat Shock Protein 90 (HSP90) Inhibitors [Number; unit: participants]
  Yes | 5
  No | 21
  Unknown | 1
Prior Systemic Treatment for GIST [Number; unit: participants]
  Yes | 27
  No | 0
Number of Prior Systemic Treatment Regimens for GIST [Mean (Standard Deviation); unit: regimens] | 5.85 (2.476)
Best Response From Prior Systemic Treatment [Number; unit: participants] — Target Lesion Response Criteria, RECIST (version 1.0)
  * Complete response - disappearance of all target lesions
  * Partial response - at least a 30% decrease in the sum of the longest diameter of target lesions
  * Stable disease - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease
  * Progressive disease - at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of 1 or more new lesions
  participants
    Complete response | 3
    Partial response | 6
    Stable Disease | 17
    Progressive disease | 1
    Unknown | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Showing Clinical Benefit Based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0
Description: Clinical benefit is defined as showing a complete response (CR), a partial response (PR) or stable disease (SD) for at least 16 weeks.
  * CR: disappearance of all target lesions and non-target lesions and no new lesions
  * PR: at least a 30% decrease in the sum of the longest diameter of target lesions, no disease progression for non-target lesions, and no new lesions
  * SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, no disease progression for non-target lesions, and no new lesions
Time Frame: Week 16 up to Week 47
Population: Full analysis set which included participants receiving at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 27
percentage of participants | 18.5

2. Secondary Outcome: Percentage of Participants Showing an Objective Response Based on RECIST Version 1.0
Description: Objective response included participants whose best response with confirmation was a complete response (CR) or partial response (PR) from first dose until progression or end of study.
  * CR: disappearance of all target lesions and non-target lesions and no new lesions
  * PR: at least a 30% decrease in the sum of the longest diameter of target lesions, no disease progression for non-target lesions, and no new lesions
Time Frame: Week 16 up to Week 47
Population: Full analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 27
percentage of participants | 0

3. Secondary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS)
Description: PFS was defined as the time from the baseline CT scan to disease progression per RECIST or death for any cause. Progressive disease (PD) was defined as
  * at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or
  * the appearance of 1 or more new lesions or
  * the unequivocal progression of existing nontarget lesions
Time Frame: Day 1 up to Week 47
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 27
months | 1.8 [1.6 to 3.5]

4. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival
Description: Overall survival was defined as the time from first dose to death or the date last known alive.
Time Frame: Day 1 up to week 97
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 27
months | 10.3 [5.8 to 13.6]

5. Secondary Outcome: Percentage of Participants Showing a Tumor Response During Cycle 1 in Selected Participants Measured by Positron Emission Tomography (PET)
Description: PET imaging was completed on selected patients only from one investigative site. Treatment phase PET and biopsy was completed on any day from Cycle 1 Day 2 through Day 10. PET imaging data were analyzed utilizing the European Organization for Research and Treatment of Cancer (EORTC) PET Study Group guidelines [Young H, Eur J Cancer, 1999]. Tumor response was considered a complete response (CR) or a partial response (PR).
Time Frame: Day 2 to Day 10
Population: Participants from one investigative site who provided consent for the PET/CT imaging.
Measure: Number; unit: percentage of participants
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 12
percentage of participants | 66.7

6. Secondary Outcome: Count of Participants With Treatment-Emergent Adverse Events (AEs)
Description: Treatment-emergent AEs were defined as AEs that occurred from the time of first dose through 30 days after the last dose of study medication. The Investigator graded the severity of AEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria:
  Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Life threatening Grade 5 = Death
  A Serious AE is defined as any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or constitutes an important medical event.
  Dose modification includes dose delay and dose reduction.
Time Frame: Day 1 up to Week 51
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Ganetespib 200 mg/m^2
Number analyzed (Participants) | 27
participants
  >=1 AE | 27
  >=1 AE with severity grade >=3 | 15
  >= 1 SAE | 10
  >=1 AE leading to dose modification | 10
  >=1 AE leading to dose interruption | 1
  >=1 AE leading to study drug discontinuation | 3
  >=1 AE with an outcome of death | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 51
Arm/Group | Ganetespib 200 mg/m^2
Serious Adverse Events (participants affected / at risk) | 10/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganetespib 200 mg/m^2 (N=27)
Anaemia (Blood and lymphatic system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Colonic fistula (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intussusception (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Amylase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lipase increased (Investigations) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Confusional state (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganetespib 200 mg/m^2 (N=27)
Anaemia (Blood and lymphatic system disorders) | 9
Lymphopenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 3
Arrhythmia superventribular (Cardiac disorders) | 1
Ear discomfort (Ear and labyrinth disorders) | 1
Eye pain (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 13
Vomiting (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 4
Abdominal pain lower (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Retching (Gastrointestinal disorders) | 2
Anal fissure (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 15
Asthenia (General disorders) | 2
Malaise (General disorders) | 2
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Early satiety (General disorders) | 1
Feeling jittery (General disorders) | 1
Influenza like illness (General disorders) | 1
Localised oedema (General disorders) | 1
Oedema (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Eye infection bacterial (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Compression fracture (Injury, poisoning and procedural complications) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Blood alkaline phosphatase increased (Investigations) | 7
Weight decreased (Investigations) | 5
Amylase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Lipase increased (Investigations) | 4
Activated partial thromboplastin time prolonged (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood albumin decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridaemia (Investigations) | 1
Hypocalcaemia (Investigations) | 1
Hypomagnesaemia (Investigations) | 1
Hypophosphataemia (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 8
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 2
Nightmare (Psychiatric disorders) | 2
Abnormal dreams (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Bladder pain (Renal and urinary disorders) | 1
Fanconi syndrome acquired (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Polymenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Eczema (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right, 60 days before submission for publication, to review disclosures and require deletion of its confidential information, excluding the study results. Public disclosure shall be delayed for up to 60 additional days in order for the Sponsor to file a patent application, if needed. Single center publications will be postponed until after disclosure of pooled data (all sites), or, for a period of 18 months from study completion/termination at all participating sites.